CLINICAL TRIAL: NCT00194038
Title: Aripiprazole in Late Life Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Martha Sajatovic, Case Western Reserve University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10864-01-L0363
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2010-01

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Geriatric Psychiatry; Aripiprazole
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Patients were continued on treatment with their existing mood stabilizing medication, and upon enrollment were initiated on aripiprazole augmentation treatment. The initial starting dose of aripiprazole was 5 mg/day, with gradual upward titration as tolerated. Initiation of new additional antipsychotic medications was not permitted during the course of the study, and antipsychotic medications prescribed at study start were tapered and discontinued by week 4 of the study if possible.
  Other Names: Abilify

SUMMARY:
The purpose of this research study is to analyze the effectiveness and tolerability of a new medication, aripiprazole (Abilify), in individuals age 50 years and older who have bipolar disorder (manic-depressive illness).

DETAILED DESCRIPTION:
While medications such as valproate (Depakote and others) and lithium are generally considered first-line agents in late life bipolar disorder, side effects are common, and many individuals with bipolar disorder continue to have symptoms in spite of medication treatment. A continuing unmet need is the availability of medications that are generally well- tolerated and effective in later life bipolar disorders.

Antipsychotic medications such as Abilify are known to be effective for related conditions such as schizophrenia and are also used by some physicians in clinical settings in combination with mood stabilizing medications (Lithium, Depakote and others) to treat symptoms of bipolar disorder. Currently Abilify is approved by the FDA to treat schizophrenia and to treat bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Must have Bipolar disorder as confirmed by the Mini Neuropsychiatric Interview (MINI)
* Must be age 50 or older
* Must have sub-optimal response to current psychotropic management including at least one of the following:

  * Behaviors and symptoms of irritability, agitation, mood liability or diminished ability to interact with others in their place of residence
  * Diminished ability to take care of basic personal needs in their place of residence due to symptoms of bipolar disorder
  * Intolerance to current psychotropic medications; and
* Must live in the Northeast Ohio area.

Exclusion Criteria:

* An unstable medical illness, or a medical illness, which in the opinion of the study investigators, is likely to affect the outcome of the study
* DSM-IV substance dependence (except nicotine or caffeine) within the past 3 months; or
* Receiving carbamazepine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure and pulse | 12 weeks
Weight | 12 weeks
Abnormal Involuntary Movement Scale (AIMS) | 12 weeks
Barnes Akathisia Scale (BAS) | 12 weeks
Simpson Angus Neurological Rating Scale (SAS) | 12 weeks
Basic serum chemistry - screening and 12/study end | 12 weeks
Complete blood count (CBC) with differential - screening and 12/study end | 12 weeks
Electrocardiogram - screening and 12/study end | 12 weeks
Young Mania Rating Scale (YMRS) - screening, baseline, and weeks 1, 2, 4, 8, and 12/study end | 12 weeks
Hamilton Depression Rating Scale (HAM-D) - screening, baseline, and weeks 1, 2, 4, 8, and 12/study end | 12 weeks
Clinical Global Impression (CGI) | 12 weeks
Global Assessment Scale (GAS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University School of Medicine

REFERENCES:
- [Result] Sajatovic M, Coconcea N, Ignacio RV, Blow FC, Hays RW, Cassidy KA, Meyer WJ. Aripiprazole therapy in 20 older adults with bipolar disorder: a 12-week, open-label trial. J Clin Psychiatry. 2008 Jan;69(1):41-6. doi: 10.4088/jcp.v69n0106. PMID 18312036